CLINICAL TRIAL: NCT06362928
Title: Safety and Effectiveness of the Akura Thrombectomy System in the Treatment of Acute Pulmonary Embolism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akura Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-60005
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Embolism Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Patients with Acute Pulmonary Embolism (Experimental): Patients undergoing mechanical thrombectomy for acute pulmonary embolism.
  Interventions: Device: ATC System

INTERVENTIONS:
Device: ATC System — The ATC System is designed to mechanically remove emboli and restore blood flow through the pulmonary arteries in patients experiencing acute PE

SUMMARY:
This study is a prospective, single-arm, non-randomized, interventional, multicenter feasibility study to evaluate the safety and effectiveness of percutaneous mechanical thrombectomy using the Akura Thrombectomy System in subjects with acute pulmonary embolism (PE).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is > 18 and < 90 years old
2. Clinical signs and symptoms consistent with acute PE
3. PE symptom duration ≤ 14 days
4. CTA evidence of proximal PE (filling defect in at least one main or lobar pulmonary artery as determined by the investigator)
5. CTA evidence of RV/LV ratio > 0.9 note: based on Investigator's interpretation of RV/LV ratio at baseline;
6. Systolic BP ≥ 90 mmHg note: initial SBP may be < 90 mmHg but ≥ 80 mmHg if the pressure recovers with volume resuscitation
7. Stable heart rate (HR) < 130 BPM prior to procedure
8. Patient is deemed medically eligible for interventional procedure(s), per investigator guidelines and clinical judgment.
9. Subject or legally authorized representative (LAR) is willing and able to provide written informed consent prior to receiving any non-standard of care protocol specific procedures

Exclusion Criteria:

1. Prior PE < 180 days from index procedure
2. Thrombolytic use < 48 hours prior to baseline CTA
3. Pulmonary hypertension with peak pulmonary artery systolic pressure (PASP) >70 mmHg by right heart catheterization
4. Vasopressor requirement after fluids to keep pressure at ≥90 mmHg
5. FiO2 requirement >40% or >6 LPM to keep oxygen saturation >90%
6. Hematocrit <28% (Note: hematocrit required within 6 hrs. of index procedure)
7. Platelets count <100,000/µL
8. eGFR <30 ml/min per 1.73 m2
9. International normalized ratio (INR) >3
10. Major trauma injury severity score (ISS) > 15
11. Presence of intracardiac lead in right ventricle or atrium placed within 6 months prior to screening assessment
12. Cardiovascular or pulmonary surgery within 7 days of index procedure
13. Actively progressing cancer treated by chemotherapeutics
14. Known bleeding diathesis or coagulation disorder
15. Left bundle branch block
16. History of severe or chronic pulmonary arterial hypertension
17. History of chronic left heart disease with left ventricular ejection fraction ≤ 30%
18. History of decompensated heart failure
19. History of underlying lung disease that is oxygen dependent
20. History of chest irradiation
21. History of heparin-induced thrombocytopenia (HIT)
22. Contraindication to systemic or therapeutic doses of anticoagulants
23. Known anaphylactic reaction to radiographic contrast agents that cannot be pretreated
24. Known residual iliac deep vein thrombosis (DVT), inferior vena cava (IVC) clot or clot in transit (right atrium and/or right ventricle).
25. CTA imaging or other evidence that suggest, in the opinion of the investigator, the Subject is not appropriate for aspiration thrombectomy intervention (e.g., inability to navigate to target location, predominantly chronic clot or non-clot embolus)
26. Life expectancy <90 days, as determined by investigator
27. Female who is pregnant or nursing
28. Current participation in another investigational drug or device treatment study Note: observational or registry studies may be permitted with Sponsor approval

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-02-15 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Effectiveness | 48 hours
  Change in RV/LV ratio post index procedure
Safety: Composite of Major Adverse Device-Related Events | 48 hours post index procedure
  Device-related major bleeding at access, device-related death, clinical deterioration, pulmonary vascular injury or cardiac injury

SECONDARY OUTCOMES:
Safety: Composite of Major Adverse Events | 30 days post index procedure
  Assessment of major adverse events through 30 day follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Univ.-Klinikum LKH Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No